CLINICAL TRIAL: NCT06135610
Title: The Impact of Social Determinants of Health in a Cohort of Patients With Penetrating Trauma Injuries Before and During the COVID-19 Pandemic
Brief Title: Social Determinants of Health in Patients With Penetrating Trauma Injuries Before and During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Kern Medical Center (Other)
Responsible Party: Principal Investigator, Amber Jones, Principal Investigator, DO, MPH, Kern Medical Center
Other Study IDs: 0001143
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Penetrating Injury; COVID-19; Social Determinants of Health
Keywords: Penetrating Trauma; Covid-19; Social Determinants of Health
MeSH Terms: conditions — Wounds, Penetrating; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-COVID: Patients identified in Kern County who presented to the emergency department with a gunshot wound (GSW), stab wound, or assault between March 2019 and February 2020 The group was further sub-classified based on the incident zip code. Kern County zip codes were combined into urban regions as NW (zip codes:93312, 93314), NE (93301, 93305, 93306, 93308), SW (93311, 93313), and SE (93304, 93307, 93309, 93241), with a separate category defined as rural (outside Bakersfield city limits).
- COVID: Patients identified in Kern County who presented to the emergency department with a gunshot wound (GSW), stab wound, or assault between March 2020 - February 2021. The group was then further sub-classified based on the incident zip code. Kern County zip codes were combined into urban regions as NW (zip codes:93312, 93314), NE (93301, 93305, 93306, 93308), SW (93311, 93313), and SE (93304, 93307, 93309, 93241), with a separate category defined as rural (outside Bakersfield city limits).
  Interventions: Diagnostic Test: Postive SAR-CoV-2 PCR nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Postive SAR-CoV-2 PCR nasopharyngeal swab — Diagnosed Covid-19 confirmed by a positive of SAR-CoV-2 PCR nasopharyngeal swab.
  Groups: COVID

SUMMARY:
Investigators report on the impact of the COVID-19 stay-at-home order concerning penetrating violence and its association within different socioeconomic regions within the county. The distribution and volume of violent offenses prior to the stay-at-home order was compared to during the stay-at-home order. This bears a crucial significance in our injury prevention and education efforts within our community.

DETAILED DESCRIPTION:
Investigators hypothesized that the COVID-19 'Stay At Home" order contributed to an increase in the incidence of violent traumatic injuries, particularly in areas with lower socioeconomic status in Kern County, as measured by census data, which was previously shown to be true in other areas of America. Investigators conducted a retrospective analysis of injuries sustained before and during the pandemic and further explored the median income of the area of injury to determine if socioeconomic status was a determinant of violent crime incidence rates. This study aims to better understand the causality of the increase in crime, further analyze the results, and identify trends in future public health crises.

This retrospective cross-sectional minimal risk study utilized the Kern Medical's trauma registry to identify patients in Kern County who presented to the emergency department with a gunshot wound (GSW), stab wound, or assault between March 2019 and February 2021. All reported blunt injuries, motor vehicle incident-related injuries, suicide attempts, or unintentional injuries were excluded. Each case was categorized as pre-COVID (March 2019 - February 2020) or COVID (March 2020 - February 2021) and further subclassified based on the incident zip code. Kern County zip codes were combined into urban regions as NW (zip codes:93312, 93314), NE (93301, 93305, 93306, 93308), SW (93311, 93313), and SE (93304, 93307, 93309, 93241), with a separate category defined as rural (outside Bakersfield city limits). These regions were also defined by median income as lower income (≤$50k: NW and SW) and higher income (>$50k: NE, SE, Rural) based on California census data. This study was approved by the Institutional Review board of Kern Medical Hospital.

Tabulated data were analyzed using odds ratios, chi-square tests of Independence, Woolf's test for homogeneity of Odds Ratios, Fisher's exact test, and the Generalized Cochran-Mantel-Haenszel test. Regions were identified with median incomes of ≤$50k and >$50K then were analyzed using a Cochran-Mantel-Haenszel test with an ad hoc analysis looking at the occurrence of GSWs and stab wounds pre-COVID and during COVID. A Bonferroni p-value adjustment was performed for all multiple comparison p-values. Additional demographic variables were collected, including patient demographics, follow-up, and death, but they were not included in these analyses.

ELIGIBILITY:
Inclusion Criteria:

* emergency department presentation with a gunshot wound (GSW), stab wound, or assault between March 2019 and February 2021.

Exclusion Criteria:

* All reported blunt injuries, motor vehicle incident-related injuries, suicide attempts, or unintentional injuries were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Kern County who presented to the emergency department with a gunshot wound (GSW), stab wound, or assault between March 2019 and February 2021. All reported blunt injuries, motor vehicle incident-related injuries, suicide attempts, or unintentional injuries were excluded. Each case was categorized as pre-COVID (March 2019 - February 2020) or COVID (March 2020 - February 2021) and further subclassified based on the incident zip code. Kern County zip codes were combined into urban regions as NW (zip codes:93312, 93314), NE (93301, 93305, 93306, 93308), SW (93311, 93313), and SE (93304, 93307, 93309, 93241), with a separate category defined as rural (outside Bakersfield city limits). These regions were also defined by median income as lower income (≤$50k: NW and SW) and higher income (>$50k: NE, SE, Rural) based on California census data.
Sampling Method: Non-Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Penetrating injury rate | March 2019 - Februrary 2021
  Penetrating injury rate including gunshot wounds, stab wounds or other penetrating assult

CONTACTS AND LOCATIONS:
Locations (1):
- Kern Medical Center, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No